CLINICAL TRIAL: NCT01289405
Title: Phonoaudiologic Therapy as an Adjunct to the Continuous Positive Airway Pressure Treatment on Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Phonoaudiologic Therapy Adjunct to Treatment on Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 2002/08
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: obstructive sleep apnea; oropharyngeal exercises; speech therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Communication Disorders | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo exercices (Placebo Comparator): relaxation exercises and stretching neck, without therapeutic purpose.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- phonoaudiologic therapy (Active Comparator): isometric and isotonic exercises to improve posture, mobility and muscle tone of the soft palate, pharyngeal constrictor muscles, tip and base of tongue, cheeks and lips.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — mechanical splint to open airway during sleep, considered the gold standard treatment for patients with obstructive sleep apnea

SUMMARY:
Objective: to evaluate the effects of a speech therapy exercises program in the treatment of Obstructive Sleep Apna Syndrome (OSAS) patients based on the clinical and polysomnography (PSG) parameters.

Methods: 80 patients with OSAS will be evaluated: men, 25-65 years old, body mass index < 35 kg/m2 and scores of Epworth Sleepiness Scale > 9. Patients will be divided into four groups: I: 20 patients with OSAS underwent speech therapy; II: 20 patients with OSAS underwent placebo therapy of Speech Therapy; III: 20 patients starting treatment with CPAP underwent speech therapy; IV: 20 patients starting treatment with CPAP without speech therapy or placebo. The speech therapy include isometric and isotonic exercises to improve posture, mobility and muscle tone of the soft palate, pharyngeal constrictor muscles, tip and base of tongue, cheeks and lips. Placebo therapy includes relaxation exercises and stretching neck, without therapeutic purpose. Both therapies are applied for three months, three times a day, lasting 20 minutes each session. During the treatment, the subjects will be monitored in weekly meetings, for orientation and description of the exercises and return of the fulfilled exercises diary. The subjects will also be followed at the CPAP clinic in returns after one week, a month and at the end of the study. Conduct assessments before and after treatment and after twenty one days washout, including: assessing the upper airway, anthropometric investigation of the facial skeleton and speech of Orofacial, questionnaires (Epworth Sleepiness Scale, FOSQ, General Segment and use of CPAP, WHOQOL-BREF, snoring), Psychomotor Vigilance Test and PSG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent diagnosis of OSAS
* Body mass index (BMI) < 35 kg/m2

Exclusion Criteria:

* Facial malformations
* Regular use of hypnotic medications
* Hypothyroidism
* Previous stroke
* Neuromuscular disease
* Heart failure
* Coronary disease
* Severe obstructive nasal disease

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
objective sleep pattern | 90 days
  sleep stages, arousals, apnea-hypopnea index, oxyhemoglobin saturation evaluated by polysomnography

SECONDARY OUTCOMES:
somnolence | 90 days
  score of Epworth Sleepiness Scale
Quality of Life | 90 days
  score of WHOQOL-BREF and FOSQ questionnaires
Cognition | 90 days
  Evaluations of Psychomotor Vigilance Test

CONTACTS AND LOCATIONS:
Overall Officials: Lia Rita A Bittencourt, MD, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Associação Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Diaferia G, Santos-Silva R, Truksinas E, Haddad FLM, Santos R, Bommarito S, Gregorio LC, Tufik S, Bittencourt L. Myofunctional therapy improves adherence to continuous positive airway pressure treatment. Sleep Breath. 2017 May;21(2):387-395. doi: 10.1007/s11325-016-1429-6. Epub 2016 Dec 2. PMID 27913971